CLINICAL TRIAL: NCT06793592
Title: Recruiting Healthcare Workers on the International Labor Market: A Megastudy
Acronym: MORE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Harvard University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BSS-2024-204-A; CF23-1514 (Other Grant/Funding Number: Carlsberg Foundation)
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: recruitment; labor migration; healthcare; megastudy
MeSH Terms: interventions — NMT1 protein, S pombe

STUDY DESIGN:
Who Masked: Participant
Masking Description: Recruiters interacting with candidates will see only the recruitment message text they are sharing but will remain unaware of specifics of the design and pre-analysis plan.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Simplified direct message without employer value proposition (Experimental): Study participants in this condition will receive the following recruitment message via LinkedIn InMail:
  Work in Denmark, FIRST NAME!
  In Denmark, there are many open positions for nurses in public healthcare facilities. As a nurse, you'll ensure patients get the care they need. You will identify patients' needs and implement and monitor their corresponding medical plan and treatment. If this sounds like a job you would like, this is the place for you.
  Read more and apply: [LINK]
  Recruiter name Talent Consultant A State of Denmark
  Interventions: Behavioral: Simplified direct message with no employer value proposition
- Family support during relocation (Experimental): Study participants in this condition will receive the following recruitment message via LinkedIn InMail:
  Work in Denmark and we will help your family with the transition, FIRST NAME!
  The process of getting started as a nurse in Denmark is easy. When you move, we will provide support for your partner to get a job and top-quality childcare and public education for your children. If you want to live in a country where your whole family will feel supported, this is the place for you.
  Read more and apply: [LINK]
  Recruiter name Talent Consultant A State of Denmark
  Interventions: Behavioral: Behaviorally informed recruitment message
- Work-life balance (Experimental): Study participants in this condition will receive the following recruitment message via LinkedIn InMail:
  Work in Denmark and enjoy work-life balance, FIRST NAME!
  In Denmark, we care for the people who care for patients, which is why work-life balance is a priority. If you want to work 37 hours a week, with six weeks of holiday and a schedule planned in advance, this is the place for you.
  Read more and apply: [LINK]
  Recruiter name Talent Consultant A State of Denmark
  Interventions: Behavioral: Behaviorally informed recruitment message
- Pay (Experimental): Study participants in this condition will receive the following recruitment message via LinkedIn InMail:
  Work in Denmark and enjoy higher pay, FIRST NAME!
  Denmark is among the highest paying countries for nurses in Europe with an average annual salary of 47,000 Euros. If you are looking for your work to be valued in terms of a higher pay, this is the place for you.
  Read more and apply: [LINK]
  Recruiter name Talent Consultant A State of Denmark
  Interventions: Behavioral: Behaviorally informed recruitment message
- Job benefits (Experimental): Study participants in this condition will receive the following recruitment message via LinkedIn InMail:
  Work in Denmark and enjoy more benefits at work, FIRST NAME!
  We will offer you several benefits at work: six weeks of paid vacation, flexible working hours planned in advance, free healthcare and retirement benefits. If you are looking for a job that rewards your commitment, this is the place for you.
  Read more and apply: [LINK]
  Recruiter name Talent Consultant A State of Denmark
  Interventions: Behavioral: Behaviorally informed recruitment message
- Livability of Denmark (Experimental): Study participants in this condition will receive the following recruitment message via LinkedIn InMail:
  Work in Denmark and enjoy a livable country, FIRST NAME!
  Denmark is top ranked in terms of livability because it outperforms other European countries in factors such as safety, trust, and life satisfaction. If you want to live in a country where quality of life is top, this is the place for you.
  Read more and apply: [LINK] Recruiter name Talent Consultant A State of Denmark
  Interventions: Behavioral: Behaviorally informed recruitment message
- Career advancement (Experimental): Study participants in this condition will receive the following recruitment message via LinkedIn InMail:
  Work in Denmark and advance your career, FIRST NAME!
  We will offer you plenty of opportunities for career development through academic diplomas or job promotions that allow for more responsibility. If you want to advance your nursing career, this is the place for you.
  Read more and apply: [LINK]
  Recruiter name Talent Consultant A State of Denmark
  Interventions: Behavioral: Behaviorally informed recruitment message
- General support during relocation (Experimental): Study participants in this condition will receive the following recruitment message via LinkedIn InMail:
  Work in Denmark and we will help you with the transition, FIRST NAME!
  The process of getting started as a nurse in Denmark is easy. We will help with finding a home, learning the language and getting settled. If you want to live in a country that will help you relocate, this is the place for you.
  Read more and apply: [LINK]
  Recruiter name Talent Consultant A State of Denmark
  Interventions: Behavioral: Behaviorally informed recruitment message
- Competent healthcare system (Experimental): Study participants in this condition will receive the following recruitment message via LinkedIn InMail:
  Work in Denmark in a well-functioning system, FIRST NAME!
  The Danish healthcare system is one of the highest ranked in Europe because of a high number of nurses and doctors. If you want to work in a country with a competent and well-functioning healthcare system, this is the place for you.
  Read more and apply: [LINK]
  Recruiter name Talent Consultant A State of Denmark
  Interventions: Behavioral: Behaviorally informed recruitment message
- Social support at work (Experimental): Study participants in this condition will receive the following recruitment message via LinkedIn InMail:
  Work in Denmark and enjoy a supportive team, FIRST NAME!
  We will offer you opportunities to work alongside a nurse partner because working in healthcare can be stressful. If you value supportive work environments, this is the place for you.
  Read more and apply: [LINK]
  Recruiter name Talent Consultant A State of Denmark
  Interventions: Behavioral: Behaviorally informed recruitment message
- Control group (no message) (Experimental): Does not receive a recruitment message
  Interventions: Behavioral: No message

INTERVENTIONS:
Behavioral: Behaviorally informed recruitment message — Study participants will receive a behaviorally informed recruitment message that highlights an employer value proposition.
  Arms: Career advancement; Competent healthcare system; Family support during relocation; General support during relocation; Job benefits; Livability of Denmark; Pay; Social support at work; Work-life balance
Behavioral: Simplified direct message with no employer value proposition — Study participants will receive a simplified message that does not highlight any specific employer value proposition.
  Arms: Simplified direct message without employer value proposition
Behavioral: No message — Study participants will not receive a recruitment message.
  Arms: Control group (no message)

SUMMARY:
Public health organizations in Denmark and most Organization for Economic Cooperation and Development (OECD) countries face an urgent demand for nursing staff. However, existing research does not yet offer a systematic understanding of how to attract talent to public healthcare organizations from the international labor markets.

In this study, the researchers will collaborate with a network of Danish public healthcare service providers led by the implementation partner Copenhagen Capacity to implement a large-scale megastudy (n=110,000), aimed at recruiting nurses and nursing assistants from across the European Union to Denmark. The study takes an employer-driven recruitment approach, co-designing and implementing a national recruitment campaign that uses social media job platforms to identify and contact potential recruits with a direct, personal message coming from a national recruitment agency.

The study aims to answer three research questions:

Research Question 1: Does receiving a behaviorally informed recruitment message (relative to a message with no employer value proposition) motivate a prospective employee to engage? Research Question 2: Does receiving any recruitment message (relative to receiving no message) motivate a prospective employee to engage? Research Question 3: What factors - that could be emphasized as employer value propositions in a short message - would motivate a prospective employee to engage?

Study participants will be randomly assigned to one of 10 treatment conditions in which they'll receive a recruitment message highlighting different employer value propositions or a simplified message including no employer value proposition, or to a control group that will receive no message.

Researchers will analyze differences across groups in terms of engagement after receiving a recruitment message, which can involve accepting, declining, responding to the message, clicking on a link within the message, and in this link registering to a national database to receive regular newsletters featuring job advertisements.

ELIGIBILITY:
We define inclusion/exclusion criteria as follows:

* Their current/primary country/location listed on the public profile corresponds to any of the 26 European Union countries (all European Union member states except Denmark), as well as Norway and Switzerland.
* They have fewer than 10 years of work experience if their profile includes job entries with corresponding start and end dates. Profiles without job dates (preventing calculation of total experience) or with no listed work experience will also be included in the sample.
* Their public profile includes any of the following terms in their job titles, either as full terms or partial matches, in English or any local language: "Nurse", "Nursing Assistant", "Registered Nurse", "Intensive Care Nurse", "Emergency Room Nurse", "Surgical Nurse", "Travel Nurse", "Nurse Practitioner", or "Nursing Student" Additionally, their education section lists any of these terms, either as full terms or partial matches: "Nurse", "Nursing", "Registered Nursing/Registered Nurse" or "Nursing Science". We exclude job titles that indicate roles outside the scope of our interest. Examples include: "Midwife", "Dental nurse", "Veterinary nurse", "Occupational health/company nurse", "Cosmetology nurse", "Military/Fire nurse", "Retired nurse", "Nurse consultant/advisor", and "Nurse teacher/professor". In addition, we drop any positions or education records where the job/degree title appears 5 or fewer times in the sample.
* Individuals with five or more connections on their LinkedIn profile.
* Individuals with an active profile (i.e. a profile that has been updated) in 2024.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110000 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Any engagement with recruitment message | Up to 4 weeks after reception of recruitment message
  A binary indicator defined at the individual level, where 1 indicates that the individual, up to 4 weeks after receiving the message, accepted or declined the recruitment message, and/or wrote a text response to the recruitment message, and/or clicked on the link within the message.

SECONDARY OUTCOMES:
Positive engagement with recruitment message | Up to 4 weeks after reception of recruitment message
  A binary indicator defined at the individual level, where 1 indicates that the individual, up to 4 weeks after receiving the message, accepted the recruitment message, and/or wrote a text response to the recruitment message, and/or clicked on the link within the message. Otherwise, the variable equals 0.
Click on the landing page | Up to 4 weeks after reception of recruitment message
  A binary indicator at the individual level, where 1 indicates that the individual clicked the link to access the recruitment landing page up to 4 weeks after receiving the recruitment message. Otherwise, the variable equals 0.
Registration to the national database | Up to 12 weeks after after receiving the recruitment message (or having been expected to receive the recruitment message had they not been assigned to the control group)
  A binary indicator at the individual level, where 1 indicates that the individual submitted their email address to sign up to the national database up to 12 weeks after receiving the recruitment message (or having been expected to receive the recruitment message had they not been assigned to the control group).
  In the event that a study participant registers to the national database prior to having received a recruitment message (or for the control group, prior to the date they would have received the recruitment message), and in all other cases, the variable equals zero.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes
To avoid inadvertently disclosing participants' sensitive personal information, we cannot provide the full megastudy data publicly. However, we will provide a reduced dataset that includes the trial arm assignment, outcome variables, covariates, and an anonymized ID representing each individual. We restrict precise geographical information (e.g., replacing postal codes with broader regional descriptions) to ensure that no combination of variables can identify a group smaller than five individuals. This approach allows researchers to reproduce our main results without risking the potential de-anonymization of participants. De-identified data and materials will be made publicly available on Open Science Framework (OSF).
Supporting Information: Study Protocol, SAP, CSR, Analytic Code

REFERENCES:
- Available data/document: More information on IPD sharing — https://osf.io/preprints/osf/6pwxe